CLINICAL TRIAL: NCT00459459
Title: Prognostic Significance of Fine-Needle Aspiration Cytology Features in Papillary Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 200704016R
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2007-04

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Fine needle aspiration of the thyroid

SUMMARY:
The purpose of this study is to investigate the relationship between prognosis and fine needle aspiration cytology character of papillary thyroid cancer.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma is the most common thyroid malignancy worldwide. The influence of clinicopathologic features on prognosis has been examined, but the relationship between cytologic features obtained by fine-needle aspiration (FNA) and prognosis has been minimally studied. We retrospectively studied the cytologic features with computerized morphometry in 83 patients with usual-type papillary thyroid cancer and followed them for more than 10 years except for one with metastasis at diagnosis. The cytologic features of FNA and recurrence of cancer were examined statistically.

ELIGIBILITY:
Inclusion Criteria:

* Papillary thyroid cancer diagnosed in NTUH from 1977 to 2000

Exclusion Criteria:

* Patient without complete medical record

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shi, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- Shyang-Rong, Shih, Dou-Liou City, Yun-Lin County, Taiwan